CLINICAL TRIAL: NCT04288817
Title: Efficacy of Cryotherapy Combined With Intralesional Tuberculin Purified Protein Derivative (PPD) Versus Interlesional Tuberculin PPD Monotherapy in the Treatment of Multiple Common Warts
Brief Title: Efficacy of Cryotherapy Combined With Intralesional Tuberculin PPD Versus Intralesional Tuberculin PPD in Treatment of Multiple Common Warts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hiba A H alshaaby, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Multiple common warts
Record Dates: First submitted 2020-02-19; First posted 2020-02-28 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Common Wart
Keywords: wart; Intralesional tuberculin PPD
MeSH Terms: conditions — Warts | interventions — Tuberculin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cryotherapy and intralesional tuberculin PPD (Active Comparator): Efficacy of cryotherapy combined with intralesional tuberculin purified protein in treatment of multiple common warts
  Interventions: Biological: Tuberculin purified protein derivative
- Intralesional tuberculin PPD (Active Comparator): Efficacy of Intralesional tuberculin purified protein deravative monotherapy in the treatment of multiple common warts
  Interventions: Biological: Tuberculin purified protein derivative

INTERVENTIONS:
Biological: Tuberculin purified protein derivative — Intralesional injection of tuberculin PPD in treatment of multiple common warts

SUMMARY:
The investigate the efficacy and safety of combined 'cryo-immuno-therapy' versus intralesional tuberculin purified protein derivative (PPD) antigen immunotherapy alone for multiple common warts

DETAILED DESCRIPTION:
Common warts are benign skin lesions caused by the human papillomavirus (HPV). The dorsal surface of the hands and fingers are the main predilection sites. Cryotherapy is frequently used to eradicate common warts via necrotic destruction of HPV-infected keratinocytes or by inducing of an effective cell-mediated immune response. However, the cure rates of cryotherapy are only around (44-47%) .

Intralesional antigen immunotherapy represents a promising therapeutic approach for the treatment of different types of warts, particularly if multiple and/or recalcitrant.

The investigate the efficacy and safety of combined 'cryo-immuno-therapy' versus intralesional tuberculin purified protein n immunotherapy alone for multiple common warts.

Although intralesional immunotherapy - compared to conventional therapeutic methods - has been generally along with better outcome, lower incidence of side effects and less recurrence, it is not still approved as a standard method of treatment in patients with wart , because the majority of available studies are open-labeled and randomized, placebo-controlled trials are very scarce.

The immune system plays an important role in the spontaneous resolution of warts. The immune mechanisms against HPV include the development of cell-mediated immune response with activation of T helper1 (Th1) lymphocytes resulting in long-term immunity . Stimulation of the immune system would clear warts in other locations, eliminating the need for the local treatment for each individual wart .

Multiple studies support the use of intralesional PPD injection as an effective and valuable treatment option due to its systemic effect, especially for patients with multiple warts, with the benefit of clearance of both treated and distant warts.

ELIGIBILITY:
Inclusion Criteria:

1. A dults older than 18 years
2. multiple (>3 warts) common warts .
3. not currently using other treatments for a wart .
4. not had relapsed at least once after treatment with any of the tissue-destructive modalities.
5. Positive tuberculin skin test.

Exclusion Criteria:

* Acute febrile illness, history of asthma, allergic skin disorders.-1 2- Pregnancy or lactation. 3- Cold-induced diseases. 4- Immunosuppression.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2021-03-01 (Estimated); Study Completion 2021-05-01 (Estimated)

PRIMARY OUTCOMES:
Size of lesions | Two months
  By decreasing in size after treatment and compare the response of the lesions tow treatment lines
Number of lesions | 4 months
  The following grading system will be used to evaluate treatment response:
  *Complete response: responders who show 100% improvement (disappearance of all warts and return to normal skin markings).
  Marked response: responders who show 76 to 99% decrease in number and/or decrease in apparent size, as assessed by a clinician and photographic evaluation also known as near-complete response.
  * Moderate response: partial responders show 25 to 75% improvement.
  * No or minimal response: less than 25% decrease in size/numbers of all warts. the study

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Awad SM, Gomaa AS, Hassan HA, Tawfik YM. Efficacy of Cryotherapy Combined With Intralesional Purified Protein Derivative (PPD) Versus Intralesional PPD Monotherapy in the Treatment of Multiple Common Warts. J Cutan Med Surg. 2023 Mar-Apr;27(2):117-125. doi: 10.1177/12034754231152224. Epub 2023 Jan 27. PMID 36705474